CLINICAL TRIAL: NCT00693589
Title: Effect of Homocysteine-lowering Therapy With Folic Acid, Vitamin B12, and Vitamin B6 on Endothelium-dependent Vasodilatation of Forearm Resistance Vessels in Patients With Coronary Heart Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Allemann, Y., MD, Cardiology, Inselspital Berne
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KEK-Nr. 115/03
Record Dates: First submitted 2008-06-05; First posted 2008-06-09 (Estimated); Last update posted 2024-11-07 (Actual); Status verified 2008-06

CONDITIONS: Cardiovascular Disease; Endothelial Dysfunction
Keywords: endothelial function; flow mediated dilatation; rosuvastatin; folic acid; B vitamins
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Folic Acid; Vitamin B 12; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- R (Active Comparator): Rosuvastatin treatment for 6 weeks and after that combined treatment with rosuvastatin and vitamin supplementation for additional 6 weeks
  Interventions: Drug: folic acid, vitamin B12 and B6 and rosuvastatin
- V (Active Comparator): Vitamin supplementation with folic acid, vitamin B12 and B6 for 6 weeks and after that combined treatment with vitamin supplementation and rosuvastatin
  Interventions: Drug: folic acid, vitamin B12 and B6 and rosuvastatin

INTERVENTIONS:
Drug: folic acid, vitamin B12 and B6 and rosuvastatin — Vitamin supplementation with folic acid 1mg/d, vitamin B12 0.4mg/d and B6 10mg/d po for 6 weeks alone vs. rosuvastatin 10mg/d for 6 weeks alone and thereafter combined treatment for 6 weeks
  Other Names: Crestor

SUMMARY:
Endothelial dysfunction is an early marker of atherosclerosis and is found in patients (pts) with coronary (CAD) and peripheral artery disease (PAD). Statin-therapy has been shown to improve endothelial function in pts with CAD or PAD by reducing LDL-cholesterol and inflammatory markers. B-group vitamin-supplements have variable been reported to have positive or neutral effects on endothelial function. Therefore, we want to compare the effect of rosuvastatin and B-group vitamin supplementation on endothelial function of the forearm resistance vessels in pts with cardiovascular disease.

DETAILED DESCRIPTION:
Study design: 36 pts with CAD or PAD are randomly assigned to either rosuvastatin 10mg/d or vitamin supplementation with folic acid 1mg, vitamin B12 0.4mg and B6 10mg/d for 6 weeks in a double-blinded design. After 6 weeks all pts receive rosuvastatin and vitamin supplementation in combination for additional 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* CAD or PAD (>50% luminal stenosis), previous myocardial infarction or bypass surgery >3 month ago
* history of percutaneous coronary intervention (PTCA or stenting)
* confirmed consent

Exclusion Criteria:

* myocardial infarction or acute coronary syndrome or bypass surgery <3 month ago
* ongoing treatment with statins
* ongoing vitamin supplementation with folic acid and B vitamins
* <18 years
* active smokers
* uncontrolled arterial hypertension
* renal insufficiency
* atrial fibrillation
* liver disease
* NYHA class >2
* familial hypercholesterolemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-01; Primary Completion 2007-02 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Flow mediated dilatation (FMD) | after 6 weeks of randomized treatment and after 6 weeks of combined treatment

SECONDARY OUTCOMES:
changes in biochemistry parameters | after 6 weeks of randomized treatment and after 6 weeks of combined treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kerstin Wustmann, MD, Study Director — Cardiology, Inselspital, University hospital Bern; Yves Allemann, MD, Study Chair — Cardiology, Inselspital, University hospital Bern